CLINICAL TRIAL: NCT06247072
Title: TRK-3 Conformance to Standards for Tonometers
Status: Completed | Type: Observational
Sponsor: Topcon Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: THQ-THINC-2023-02
Record Dates: First submitted 2024-01-30; First posted 2024-02-07 (Actual); Last update posted 2024-04-08 (Actual); Status verified 2024-04

CONDITIONS: Glaucoma
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (3):
- low IOP: having low IOP in one eye
  Interventions: Device: Tonometer
- intermediate IOP: having intermediate IOP in one eye
  Interventions: Device: Tonometer
- high IOP: having high IOP in one eye
  Interventions: Device: Tonometer

INTERVENTIONS:
Device: Tonometer — measures IOP

SUMMARY:
To collect measurements of a new tonometer and show conformance to standards for tonometers.

ELIGIBILITY:
Inclusion Criteria:

1. Age at least 22 years at the time of the informed consent
2. Provide voluntary written consent for participation in the study

Exclusion Criteria:

1. Have only one functional eye
2. Have difficulty in ocular fixation or eccentric fixation in either eye
3. Have corneal scar or have a history of corneal surgery such as corneal laser surgery (cataract surgery is acceptable)
4. Have microphthalmia
5. Have buphthalmos
6. Wear contact lens (have used soft contact lenses within the last 3 months and/or hard contact lenses within the last 6 months)
7. Have dry eyes and taking prescription medication or using artificial tears daily
8. Have blepharospasm
9. Have nystagmus
10. Have keratoconus
11. Have corneal or conjunctival lesions or infections
12. Have a central corneal thickness of <500μm or >600μm
13. Have corneal astigmatism >3D
14. Have known allergy to ophthalmic anesthetics
15. Have known allergy to sodium fluorescein

Min Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Eyes with different range of IOP
Sampling Method: Non-Probability Sample
Enrollment: 125 (Actual)
Dates: Start 2024-02-02 (Actual); Primary Completion 2024-04-04 (Actual); Study Completion 2024-04-04 (Actual)

PRIMARY OUTCOMES:
IOP | 1 day
  pressure inside the eye

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - New View Optometric Center, La Mesa, California
  - Illinois College of Optometry, Chicago, Illinois

IPD SHARING:
Plan to Share IPD: No